CLINICAL TRIAL: NCT04306289
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Pain Associated With Diabetic Neuropathy
Brief Title: tDCS and Pain Associated With Diabetic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Mohammad Alwardat, postdoctoral fellowship, University of Rome Tor Vergata
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: University of Rome Tor Vergata
Record Dates: First submitted 2020-03-03; First posted 2020-03-12 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Neuropathies; Chronic Pain
Keywords: chronic pain; transcranial direct current stimulation; Diabetic Neuropathy; Quality of life
MeSH Terms: conditions — Diabetic Neuropathies; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Active Comparator): The participant will receive anodal tDCS for 20 min at an intensity of 2 mA while seated comfortably and quietly in a room. The intensity will start at 0 mA and will be incrementally increased to 2mA over the initial 30 seconds. At the 19:30 minute time point, the current will gradually be reduced from 2 mA to 0 mA.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Identical to the real tDCS, except the participants will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 for the remainder of the 20 minutes.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a noninvasive technique of neuronal modulation that has been used in different neurological conditions, neuropathic pain.

SUMMARY:
The purpose of this study is to investigate the effects of anodal transcranial direct current stimulation (tDCS) on pain intensity associated with diabetic neuropathy. The investigators will conduct real tDCS or sham, over the left dorsolateral prefrontal cortex (DLPFC) during 6 separated days. They will evaluate pain intensity, sleep quality, quality of life and anxiety and depression symptoms via clinical validated scales.

The research question is whether tDCS can lessen neuropathic pain and improve sleep, psychological status and quality of life in patients with diabetic neuropathy.

It is hypothesized, that less neuropathic pain and improved sleep, psychological status and quality of life after the tDCS sessions.

DETAILED DESCRIPTION:
Background: Worldwide, the prevalence of diabetes mellitus (DM) and its chronic complications are reaching epidemic proportions. By 2045 DM expected to affect 629 million persons. Diabetic neuropathy is one of the most common complications of DM and is actually the set of heterogeneous clinical forms. Among diabetic neuropathies, generalized, focal or multifocal forms are distinguished. The most typical and most common form (up to 80% of cases is sensory-motor polyneuropathy. It has recently been redefined as a length-dependent symmetric sensory-motor polyneuropathy attributable to metabolic and microvascular alterations following exposure to chronic hyperglycemia and cardiovascular risk cofactors. Painful diabetic peripheral neuropathy (PDPN) may be considered a variant; about 15-25% of patients have painful diabetic polyneuropathy.

According to the definition of neuropathic pain of the International Association for the Study of Pain (IASP), PDPN is considered as asymmetric sensory-motor polyneuropathy chronic in which neuropathic pain has been present, for at least 3 months, as direct consequence abnormalities of the peripheral somatic-sensitive system following diabetic pathology. Sensory symptoms are more evident than motor symptoms; which is appear in the most distal portions of the limbs and progress proximally according to a "glove" or "sock" distribution associated with paresthesias and dysesthesias. The clinical symptoms are related to the type of nerve fiber involved and typically there are "positive" (tingling, burning, pain, allodynia) or "negative" sensory symptoms (loss of sensitivity, numbness). The involvement of small sensitive fibers causes a reduction in thermal sensitivity and pain and this, in turn, contributes to the deficits in tactile and proprioceptive sensitivity to increase the risk of a foot injury.

The PDPN is associated with negative repercussions on the quality of life (QoL), activities of daily livings, sleep disorders, and is the major determinant of depressive symptoms in patients with PDNP. In fact, depression and sleep disturbances play a negative prognostic role in the general and diabetic population, and sleep disturbances are associated with glycated hemoglobin levels higher than 0.35% in type 2 diabetes. The presence of PDPN determines an increase in the use of medical care and social costs, both directly related to treatments, and indirect secondary to the reduction of working capacity. The presence of chronic pain of any nature increases the risk of difficulties in the self-management of diabetes, in relation to taking therapy, physical activity, adherence to the diet, foot care and even glycemic self-monitoring.

Transcranial Direct Current Stimulation (tDCS) has shown promising results for the treatment of chronic pain in several types of diseases, being a good and non-invasive alternative to treat pain in PDPN patients. Also, based on studies that showed changes in the brain activity of chronic pain patients and on the difficulties faced to treat PDPN, there is a need to conduct clinical trials using new techniques, such as neuromodulation, to help these patients to control their pain. Therefore, tDCS emerges as a new tool to be coupled with other effective treatments already used for these patients.

The dorsolateral prefrontal cortex (DLPFC) is a functionally and structurally heterogeneous region as well as a key area of numerous brain networks involved in the processing of cognition effect. Numerous studies have shown that some chronic pain syndromes are associated with a reduction in the volume of the gray matter of DLPFC. Some studies show that pain relief manages to reverse these structural changes PDPN. Moreover, previous studies reported that DLPFC stimulation induces a significant analgesic and antidepressant effect.

Hypothesis: The investigators believe that neuromodulation by tDCS over the left DLPFC would decrease the pain intensity and improve the general quality of life in patients with PDPN.

Objectives: general PURPOSE Investigate if anodal tDCS over left DLPFC has analgesic effects in patients with PDPN.

Specifics purposes 1- Evaluate the tDCS effects over pain intensity; 2- Evaluate if tDCS has any effect on sleep quality, depression, anxiety, and quality of life.

Randomization: The subjects will be allocated consecutively to randomization as an intervention order using the tool from the randomization.com website (Dallal GE, http://www.randomization.com). The investigators will use the second generation suggested for crossover studies.

Data Collection Procedure: All subjects will be treated using two different interventions (groups respecting the washout period of six weeks to avoid residual effects. The intervention order will be determined by randomization per group of interventions. Subjects will be contacted by phone and asked if they want to participate in the study. Those who wish to participate and qualify according to the selection criteria after completing the pre-screening questionnaire will be scheduled after reading and signing the consent form (2 copies). During the second visit, all clinical and neurological assessments will be performed before and after tDCS stimulation phase. Each patient will be clinically and neurologically assessed before and after the stimulation, allowing data to be collected 4 times (T0, T1, T2, and T3).

tDCS protocol: Group Real tDCS: The participant will receive anodal tDCS over the left DLPFC and the reference electrode will place over the right forearm. The stimulation intensity will be 2mA DC delivered for 20 min (30 s step-up ramp, 30 s step-down ramp), repeated six times, during two weeks (Mon, Wed, Frid).

Group sham tDCS: Identical to the real tDCS, except the participants will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 for the remainder of the 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with painful diabetic peripheral neuropathy (PDPN) components with DN4 score ≥ 4/10, and chronic pain with an intensity of at least VAS> 4/10.
* Onset of neuropathic PDPN pain for at least 6 months.
* Pain intensity as measured by VAS> 4/10 in the week preceding inclusion in the study.
* drug-resistant patients who have no pain reduction of 50% or an improvement of at least 2 points in the Patient Global Impression of Change, having used all the classes of drugs indicated as a first, second or third line.
* Absence of glycemic de-compensation with HbA1c values <9% in the previous 6 months.
* Stability of glycemic control with changes in HbA1c in the last 6 months of less than 2%.

Exclusion Criteria

* Neurological comorbidities.
* Presence of contraindications to the use of electrotherapy (pacemaker, epilepsy, etc ...).
* Pregnancy.
* Previous neurosurgical interventions.
* psychiatric conditions.
* Cognitive impairments ( Mini-Mental Status exam (MMSE) <24).
* Presence of red flags for pain: tumors, spine fractures, non-neuropathic pain difficult to distinguish from that of the PDPN, neuropathic pain from a cause other than the PDPN.
* Severe comorbidities such as advanced renal failure, heart failure, respiratory failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-06 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain severity | Measured at baseline and immediately after the intervention
  Changes in Pain severity will be measured by Brief Pain Inventory (BPI) to determine the effect of anodal Transcranial direct current stimulation (tDCS) in reducing pain of subjects with pain associated with diabetic neuropathy.

SECONDARY OUTCOMES:
Changes in Depression severity | Measured at baseline and immediately after the intervention
  Changes in depression severity will be measured by Hamilton Depression scale (HAM-D) to determine the effect of anodal Transcranial direct current stimulation (tDCS) in reducing depression severity of subjects with pain associated with diabetic neuropathy.
Changes in Anxiety severity | Measured at baseline and immediately after the intervention
  Changes in Anxiety severity will be measured by Hamilton Anxiety scale (HAM-A) to determine the effect of anodal Transcranial direct current stimulation (tDCS) in reducing anxiety severity of subjects with pain associated with diabetic neuropathy.
Changes in sleep quality | Measured at baseline and immediately after the intervention
  Changes in Sleep quality will be measured by Pittsburgh sleep quality index (PSQI) to determine the effect of anodal Transcranial direct current stimulation (tDCS) in improving sleep quality of subjects with pain associated with diabetic neuropathy.
Changes in Quality of Life | Measured at baseline and immediately after the intervention
  Changes in quality of life will be measured by SF-36 to determine the effect of anodal Transcranial direct current stimulation (tDCS) in improving quality of life of subjects with pain associated with diabetic neuropathy.
Changes in Pain related to disability | Measured at baseline and immediately after the intervention
  The investigators will use the Pain Disability Index (PDI) to assess changes in pain related to disability.
Changes in Pain Catastrophizing | Measured at baseline and immediately after the intervention
  The investigators will use the Pain Catastrophizing Scale (PCS) to assess changes in pain Catastrophizing.
Changes in Neuropathic Pain Symptom | Measured at baseline and immediately after the intervention
  Changes in neuropathic pain symptoms will be measured by Neuropathic Pain Symptom Inventory (NPSI) to determine the effect of anodal Transcranial direct current stimulation (tDCS) in improving and/or reducing neuropathic pain symptom of subjects with pain associated with diabetic neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Slivia Natoli, MD, PhD, Study Director — Department of Clinical Science and Translational Medicine, University of Rome Tor Vergata, 00133 Rome, Italy.
Locations (1):
- Prof. Silvia Natoli, Rome, Lazio, Italy

REFERENCES:
- [Background] Dyck PJ, Kratz KM, Karnes JL, Litchy WJ, Klein R, Pach JM, Wilson DM, O'Brien PC, Melton LJ 3rd, Service FJ. The prevalence by staged severity of various types of diabetic neuropathy, retinopathy, and nephropathy in a population-based cohort: the Rochester Diabetic Neuropathy Study. Neurology. 1993 Apr;43(4):817-24. doi: 10.1212/wnl.43.4.817. PMID 8469345
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Tesfaye S, Chaturvedi N, Eaton SE, Ward JD, Manes C, Ionescu-Tirgoviste C, Witte DR, Fuller JH; EURODIAB Prospective Complications Study Group. Vascular risk factors and diabetic neuropathy. N Engl J Med. 2005 Jan 27;352(4):341-50. doi: 10.1056/NEJMoa032782. PMID 15673800
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Daousi C, MacFarlane IA, Woodward A, Nurmikko TJ, Bundred PE, Benbow SJ. Chronic painful peripheral neuropathy in an urban community: a controlled comparison of people with and without diabetes. Diabet Med. 2004 Sep;21(9):976-82. doi: 10.1111/j.1464-5491.2004.01271.x. PMID 15317601
- [Background] Abbott CA, Malik RA, van Ross ER, Kulkarni J, Boulton AJ. Prevalence and characteristics of painful diabetic neuropathy in a large community-based diabetic population in the U.K. Diabetes Care. 2011 Oct;34(10):2220-4. doi: 10.2337/dc11-1108. Epub 2011 Aug 18. PMID 21852677
- [Background] Alleman CJ, Westerhout KY, Hensen M, Chambers C, Stoker M, Long S, van Nooten FE. Humanistic and economic burden of painful diabetic peripheral neuropathy in Europe: A review of the literature. Diabetes Res Clin Pract. 2015 Aug;109(2):215-25. doi: 10.1016/j.diabres.2015.04.031. Epub 2015 May 6. PMID 26008721
- [Background] Binns-Hall O, Selvarajah D, Sanger D, Walker J, Scott A, Tesfaye S. One-stop microvascular screening service: an effective model for the early detection of diabetic peripheral neuropathy and the high-risk foot. Diabet Med. 2018 Jul;35(7):887-894. doi: 10.1111/dme.13630. Epub 2018 May 10. PMID 29608799
- [Background] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Background] D'Amato C, Morganti R, Greco C, Di Gennaro F, Cacciotti L, Longo S, Mataluni G, Lauro D, Marfia GA, Spallone V. Diabetic peripheral neuropathic pain is a stronger predictor of depression than other diabetic complications and comorbidities. Diab Vasc Dis Res. 2016 Nov;13(6):418-428. doi: 10.1177/1479164116653240. Epub 2016 Jun 22. PMID 27334483
- [Background] Ziegler D, Rathmann W, Dickhaus T, Meisinger C, Mielck A; KORA Study Group. Neuropathic pain in diabetes, prediabetes and normal glucose tolerance: the MONICA/KORA Augsburg Surveys S2 and S3. Pain Med. 2009 Mar;10(2):393-400. doi: 10.1111/j.1526-4637.2008.00555.x. Epub 2009 Jan 16. PMID 19207236
- [Background] Van Acker K, Bouhassira D, De Bacquer D, Weiss S, Matthys K, Raemen H, Mathieu C, Colin IM. Prevalence and impact on quality of life of peripheral neuropathy with or without neuropathic pain in type 1 and type 2 diabetic patients attending hospital outpatients clinics. Diabetes Metab. 2009 Jun;35(3):206-13. doi: 10.1016/j.diabet.2008.11.004. Epub 2009 Mar 17. PMID 19297223
- [Background] Wu YJ, Lin CC, Yeh CM, Chien ME, Tsao MC, Tseng P, Huang CW, Hsu KS. Repeated transcranial direct current stimulation improves cognitive dysfunction and synaptic plasticity deficit in the prefrontal cortex of streptozotocin-induced diabetic rats. Brain Stimul. 2017 Nov-Dec;10(6):1079-1087. doi: 10.1016/j.brs.2017.08.007. Epub 2017 Aug 24. PMID 28870510
- [Background] Kim YJ, Ku J, Kim HJ, Im DJ, Lee HS, Han KA, Kang YJ. Randomized, sham controlled trial of transcranial direct current stimulation for painful diabetic polyneuropathy. Ann Rehabil Med. 2013 Dec;37(6):766-76. doi: 10.5535/arm.2013.37.6.766. Epub 2013 Dec 23. PMID 24466511
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120